CLINICAL TRIAL: NCT06113744
Title: A Randomised, Blinded, Parallel-controlled Phase 1 Clinical Trial to Evaluate the Safety and Preliminary Immunogenicity of a COVID-19 mRNA Vaccine in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety and Immunogenicity of COVID-19 Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Collaborators: Shulan (Hangzhou) Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZSVG-02-O-2022-P1
Record Dates: First submitted 2023-10-31; First posted 2023-11-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Low-dose test vaccine, 1 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 10 μg
- Mid-dose test vaccine, 1 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 30 μg
- High-dose test vaccine, 1 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 60 μg
- Placebo, 1 dose (Placebo Comparator)
  Interventions: Biological: Placebo
- Low-dose test vaccine, 2 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 10 μg
- Mid-dose test vaccine, 2 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 30 μg
- High-dose test vaccine, 2 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 60 μg
- Placebo, 2 doses (Placebo Comparator)
  Interventions: Biological: Placebo
- Active control vaccine, 2 doses (Active Comparator)
  Interventions: Biological: COVID-19 Vaccine (Vero Cell) ,Inactivated

INTERVENTIONS:
Biological: Placebo — saline
  Arms: Placebo, 1 dose; Placebo, 2 doses
Biological: COVID-19 Vaccine (Vero Cell) ,Inactivated — COVILO
  Arms: Active control vaccine, 2 doses
Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 10 μg — Low-dose
  Arms: Low-dose test vaccine, 1 dose; Low-dose test vaccine, 2 dose
Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 30 μg — Mid-dose
  Arms: Mid-dose test vaccine, 1 dose; Mid-dose test vaccine, 2 dose
Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) 60 μg — High-dose
  Arms: High-dose test vaccine, 1 dose; High-dose test vaccine, 2 dose

SUMMARY:
A randomised, blinded, parallel-controlled phase 1 clinical trial to evaluate the safety and preliminary immunogenicity of a COVID-19 mRNA vaccine in a healthy population aged 18 years and older, and to investigate immunisation doses.

DETAILED DESCRIPTION:
The phase 1 clinical trial is conducted in a randomised, blinded, parallel-controlled design to assess the safety, immunogenicity and immune persistence. Subjects will be divided into two age groups (18-59 and ≧60 years of age), and within the groups, subjects will be subdivided into three dose groups (10 μg,30 μg and 60 μg). The immunisation procedure is divided into one-dose group and two-dose group (0, 28 days).

The total sample size is 164 subjects. 12 subjects will be assigned to each group according to different age, dose and immunisation procedure, respectively. In addition, 20 subjects (10 aged 18-59 years and 10 aged ≧60 years) will be enrolled as active control and vaccinated with 2 doses of inactivated Covid vaccine (Vero cell) (0, 28 days).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged ≥18 years of age;
2. Subjects who are in good physical condition as judged by the investigator based on medical history, physical examination and clinical laboratory tests;
3. Subjects who have not been previously vaccinated with a Covid-19 vaccine or who have received the last dose (total dose ≤ 3 doses) of a Covid-19 vaccine at least 6 months ago;
4. Subjects who have not been previously infected with Covid-19, or whose nucleic acid or antigen test has turned negative for more than 1 month after previous Covid-19 infection;
5. Subjects who have used effective contraception since 2 weeks prior to enrolment;
6. Subjects or their delegates are able to understand the study procedures, have provide written informed consent, and are able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

1. Females of childbearing potential who have a positive pregnancy test, are pregnant, breastfeeding, or planning to become pregnant within 12 months; males: whose spouse is planning to become pregnant within 1 year;
2. History of epilepsy, convulsions or seizures, psychosis or family history of psychosis;
3. Subjects who were using antipyretic, analgesic or anti-allergic drugs within 3 days before enrolment;
4. Have a previous history of severe allergy to any medication or vaccination (e.g. acute allergic reaction, urticaria, skin eczema, dyspnoea, angioneurotic oedema, or abdominal pain) or allergy to known components of a Covid-19 vaccine;
5. Have a history of hospital-diagnosed thrombocytopenia or other coagulation disorders;
6. Have a history of hospital-diagnosed known immunological impairment or hypofunction;
7. Subjects who have received immunoenhancement or immunosuppressant therapy (continuous use by oral or infusion for more than 14 days) within 3 months, and whole blood, plasma, or immunoglobulin within 1 month;
8. Known or suspected concomitant serious diseases, including: respiratory diseases, acute infections or active chronic diseases, liver and kidney diseases, severe diabetes, malignant tumours, infectious or allergic skin diseases, cardiovascular disease, and HIV infection (with test report);
9. Subjects suffering from various acute diseases or in the acute exacerbation of chronic diseases within 3 days before vaccination;
10. Subjects with clinically significant abnormalities in blood biochemistry, blood routine, urine routine, coagulation function, thyroid function, and myocarditis-related indicators detected during the screening;
11. Received live attenuated vaccine within 1 month before vaccination;
12. Received inactivated vaccine within 14 days before vaccination;
13. Axillary temperature ≥37.3℃;
14. Who have participated in other clinical trials within 3 months prior to the first dose of vaccination or plan to participate in other clinical trials during the study period;
15. Other conditions that the investigator deems inappropriate for participation in this clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number and frequency of adverse event (AE) | Day 0~Day 28 after each dose of vaccination
  Incidence of local/systemic adverse reactions/events 0-14 days and 15-28 days after each dose of vaccination, and incidence of solicited adverse events within 14 days after each dose of vaccination

SECONDARY OUTCOMES:
Number and frequency of serious adverse event (SAE) | From the first dose of immunisation to 12 months after full immunisation
  Incidence of SAE from the first dose up to 12 months after full immunisation
4-fold increasing rate, geometric mean titre (GMT) and geometric mean increase (GMI) of neutralizing antibodies (Nabs) against SARS-CoV-2 on 14 days and 28 days after full immunisation | From the first dose of immunisation to 28 days after full immunisation
  4-fold increasing rate, GMT and GMI of neutralizing antibody (Nabs) against SARS-CoV-2 on 14 days and 28 days after full immunisation
Cross-neutralisation against different SARS-CoV-2 variants | From the first dose of immunisation to 28 days after full immunisation
  The cross-neutralization effect of the mRNA vaccine (Omicron strain) against different SARS-CoV-2 variants (ancestral strain, Omicron strain and main circulating strain)
4-fold increasing rate, GMT and GMI of NAbs against SARS-CoV-2 on 90, 180 and 360 days after full immunisation | Day 90~Day 360 after full immunisation
  4-fold increasing rate, GMT and GMI of NAbs against SARS-CoV-2 on 90, 180 and 360 days after full immunisation

OTHER OUTCOMES:
Changes in cytokine levels in Th1/Th2 cells induced by S protein | From before the first dose of immunisation to 28 days after full immunisation
  Cytokine (IFN-γ, IL-4, IL-2) levels in Th1/Th2 cells changed from pre-dose to 28 days after the full immunisation

CONTACTS AND LOCATIONS:
Overall Officials: Yunkai Yang, Study Chair — China National Biotec Group Company Limited
Locations (1):
- Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang, China